CLINICAL TRIAL: NCT06667648
Title: Effect of Wet Cupping Versus Moderate Intensity Aerobic Exercise on Inflammatory Markers in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, associate professor of pharmaceutics and clinical pharmacy, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy 2024
Record Dates: First submitted 2024-10-16; First posted 2024-10-31 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
Keywords: diabetes, cupping, aerobic excercise
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (No Intervention): ) attended the program of walking on a treadmill machine for eight weeks according to the following parameters: -
  * Mode of exercise: aerobic exercise.
  * Intensity: according to heart rate (60-75% of maximum heart rate) MHR=220-age.
  * Heart rate: determined by the sensor of a treadmill.
  * Duration: 40-50 min per session. Each session consisted of 5-10 minutes of warming up exercise on a treadmill without increasing speed or intensity and the same for the cooling down phase
- Group (B) (Other): Each cupping session takes about 30-40 min and can be conducted in five steps. The first step includes primary suction. In this phase, the therapist allocates specific points or areas for cupping and disinfects the area, which located at the upper back (opposite to C7), Para spinal and below scapula. A cup with a suitable size is placed on the selected site and sucked the air inside the cup by manual suction. Then the cup was applied to the skin and left for a period of 3 to 5 min. The second step is about puncturing. Puncturing with a needle to get out of blood the third step is about suction and bloodletting. The cup is placed back on the skin using the similar procedure described above for 3 to 5 min. The fourth step includes the removal of the cup, followed by the fifth step which includes dressing the area after cleaning and disinfecting with FDA-approved skin disinfectant.
  Interventions: Procedure: cupping session

INTERVENTIONS:
Procedure: cupping session — Each cupping session takes about 30-40 min and can be conducted in five steps. The first step includes primary suction. In this phase, the therapist allocates specific points or areas for cupping and disinfects the area, which located at the upper back (opposite to C7), Para spinal and below scapula. A cup with a suitable size is placed on the selected site and sucked the air inside the cup by manual suction. Then the cup was applied to the skin and left for a period of 3 to 5 min. The second step is about puncturing. Puncturing with a needle to get out of blood the third step is about suction and bloodletting. The cup is placed back on the skin using the similar procedure described above for 3 to 5 min. The fourth step includes the removal of the cup, followed by the fifth step which includes dressing the area after cleaning and disinfecting with FDA-approved skin disinfectant.
  Arms: Group (B)

SUMMARY:
Among all pro-inflammatory biomarkers, TNF-α first recognized to be involved in the pathenogenesis of insulin resistance, and glucose-related abnormalities that link to T2DM. TNF-α plays a vital role in the overall pathophysiology of insulin resistance especially in males with greater body mass index as compared to that in the females This trial aims to investigate the effect of wet cupping therapy versus moderate intensity aerobic exercise on inflammatory markers in diabetic patients

DETAILED DESCRIPTION:
Cupping therapy is a traditional treatment used to create suction on the skin over a painful area or acupuncture point using a bamboo or glass cup. Aerobic exercise (also known as endurance activities, cardio, or cardio-respiratory exercise) is physical exercise of low to high intensity that depends primarily on the aerobic energy-generating process. Chronic inflammation, including elevated levels of interleukin 6 (IL-6), is associated with diabetes, cardiovascular disease, and chronic kidney disease, as well as related diseases such as nonalcoholic hepatosteatosis. Amongst other triggers, elevated IL-6 levels may arise due to excess adipose tissue and can cause, for example, aberrant glucose metabolism leading to diabetes and other manifestations of the ensuing glucotoxicity in many tissues and organs, including the vasculature and other parts of the heart and the kidneys, as well as in the liver. The purpose of this study was to investigate the effect of wet cupping therapy versus moderate-intensity aerobic exercise on inflammatory markers in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* had diabetes more than 10 years ago
* body mass index of 25 to 29.9 Kg/m2

Exclusion Criteria:

* Hepatic diseases, Cancer patients, Renal failure patients, Orthopedic problems or fractures of extremities, hypertensive patients, and Neurological problems

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
interleukin 6 concentrations | 6 months
  Kits for blood sample to detect serum interleukin 6
blood sugar level mg/dl | 6 months
  blood sample to determine blood sugar level
tumor necrosis factor percent | 6 months
  kits to determine tumor necrosis factor alpha

IPD SHARING:
Plan to Share IPD: Undecided